CLINICAL TRIAL: NCT07396428
Title: Effectiveness and Implementation of a National Guideline for Acute Respiratory Tract Infections to Reduce Antibiotic Prescribing in Swiss Primary Care: the ImpProGUIDE Hybrid Type II Effectiveness-implementation Trial
Brief Title: Effectiveness and Implementation of a National Guideline for Acute Respiratory Tract Infections to Reduce Antibiotic Prescribing in Swiss Primary Care
Acronym: ImpProGUIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Collaborators: University of Zurich, Institute for Implementation Science in Health care (Unknown); Anresis, Swiss Centre for Antibiotic Resistance, University of Bern, Switzerland (Unknown); CHUV, Lausanne University Hospitals, Switzerland (Unknown); Swiss Pharmacy Association, pharmaSuisse (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Req-2024-00897; 212429 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-11-18; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Infection; Influenza-like Illness
Keywords: family medicine; primary care; implementation; hybrid design; effectiveness-implementation study; general medicine; outpatient; antibiotics; antibiotic prescribing; antimicrobial resistance; antimicrobial stewardship; guidelines; shared decision making; CRP; c-reactive protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute respiratory infection guideline implementation (Experimental): Quality circles (QC) and walk-in clinics randomized to the intervention arm will receive an overarching multifaceted implementation strategy for the new acute respiratory infection (ARI) guidelines. This includes educational materials to help the QC moderators or the person responsible for education in the clinic to lead a thematic session in autumn 2025, focusing on the use of a syndromic approach, targeted C-reactive protein (CRP) testing when bacterial infection is suspected, and shared decision-making with patients. Other facets include an information sheet and pocket card for physicians, and patient leaflets on acute cough.
  Interventions: Behavioral: Training Session on acute respiratory infection guideline within a multifaceted implementation strategy
- Usual care (No Intervention): QCs and walk-in clinics randomized to the control arm will continue their routine activities without receiving the educational materials on the new guidelines during the initial phase. In the summer 2026, these groups will be offered the same training materials provided to the intervention arm, with the option to use them in their QC sessions or internal training.

INTERVENTIONS:
Behavioral: Training Session on acute respiratory infection guideline within a multifaceted implementation strategy — Implementation strategies are deployed within quality circles, consisting of a structured educational session including a PowerPoint presentation, a facilitation guide, clinical vignettes, and printed materials for physicians and patients. The session is designed to support clinical decision-making about antibiotic use for ARI, based on targeted use of CRP and shared decision-making.
  Arms: Acute respiratory infection guideline implementation

SUMMARY:
The ImpProGUIDE study aims to find out whether implementing new Swiss national guidelines for acute respiratory infections (ARI) can help to reduce antibiotic prescribing in primary care. In Switzerland, most antibiotics are prescribed in outpatient care, and many of these prescriptions may not be needed - especially when infections are caused by viruses, which antibiotics do not treat. Reducing overuse of antibiotics is important to slow the spread of antibiotic resistance.

The new guidelines were developed by the Swiss Society for Infectious Diseases (SSI) to support family doctors in managing ARIs, based on a syndromic approach. They recommend the targeted use of point-of-care C-reactive protein (CRP) testing when bacterial infection is suspected, as well as shared decision-making with patients.

This study will be carried out in quality circles (QCs) - small groups of family doctors who meet regularly to discuss and improve clinical practice - and in walk-in clinics in French- and Italian-speaking regions of Switzerland. Each will be randomly assigned to either an "intervention" group or a "control" group.

In the intervention group, QC moderators and medical center directors will receive implementation resources to lead a session and distribute materials to their group in autumn 2025 on the new guidelines. Doctors can then decide whether or not to use the recommendations in their consultations.

In the control group, QCs and centers will continue their regular activities. They will receive access to the same educational materials later, in summer 2026.

Throughout the study, the researchers will collect de-identified data from health insurance billing records to track antibiotic prescribing and the use of diagnostic tests. Doctors and QC moderators will also be invited to complete short online surveys twice a year (10-15 minutes) and may be asked to join optional interviews or group discussions after the winter season.

The study will also explore the effectiveness of the implementation strategies on the adoption of the SSI guidelines, as well as the barriers and facilitators to adoption. This study type is known as a hybrid effectiveness implementation study, simultaneously evaluating an intervention's impact on antibiotic prescribing and the strategies used to implement the new national guidelines in a real-world setting.

Participation in the study is voluntary. Doctors can withdraw at any time. All data will be handled confidentially and in line with Swiss data protection laws.

The study is funded by the Swiss National Science Foundation. No support is received from pharmaceutical companies or manufacturers of diagnostic tests.

ELIGIBILITY:
Inclusion criteria for quality circles (QCs)

* Willing to participate in a study mainly conducted in French
* Agreeing to participate in evaluation surveys

Exclusion criteria for QCs*

- Not having any physician included in the study

Inclusion criteria for walk-in clinics

* The clinic offers general practice/primary care medicine consultations, including emergencies
* The clinic includes at least five physicians
* The clinic has an "Admission to practice charged to Swiss compulsory health insurance"
* The clinic plans to still be active in April 2026
* Located in one of the following cantons: Vaud, Geneva, Valais, Fribourg, Jura, Neuchatel, Bern, Ticino.
* Serving mainly adult patients
* Willing to participate in the study

Physicians in QCs fulfilling all of the following inclusion criteria are eligible for the study:

* Registered primary care physicians
* Specialist title in general internal medicine or practicing physician.
* Practicing in one of the following cantons: Vaud, Geneva, Valais, Fribourg, Jura, Neuchatel, Bern, Ticino.
* Participating in a QC or working in an outpatient clinic participating in the study*.
* Willing to participate in a study mainly conducted in French.
* Agreeing to participate in evaluation surveys and agreeing to be invited to interviews

Eligibility criteria for physicians in clinics :

- Having a clinical activity as primary care physician or supervising clinical activity of physicians in post-graduate training within a clinic included in the study

The only exclusion criterion for physicians is planning to retire before April 2026.

*Note: not all physicians from a QC or a clinic are expected or required to participate individually in the study, but at least one should participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Defined daily doses of antibiotics commonly used for acute respiratory infections per 1000 consultations | Over the influenza-like illness (ILI) season (6 months).
  Defined daily doses (DDD) of selected antibiotics (amoxicillin, co-amoxicillin, clarithromycin, azithromycin) per 1000 consultations, based on de-identified health insurance billing data. These antibiotics represent those most commonly prescribed for pneumonia, acute bronchitis, and upper respiratory tract infections (excluding pharyngitis, sinusitis, and otitis media).
Penetration of acute respiratory infection guidelines | Baseline and after 6 months.
  Percentage of physicians who self-declare adoption of the new acute respiratory infection (ARI) guidelines (i.e., treating patients according to the guidelines).

SECONDARY OUTCOMES:
Monthly antibiotic prescribing rate | Monthly for 12 months.
  Monthly prescribing rates expressed as: (1) DDD of antibiotics commonly used for ARI per 1000 consultations, and (2) DDD of total antibiotics per 1000 consultations.
Model-estimated differences in antibiotic use | Over the ILI season (6 months).
  Multilevel regression coefficients estimating differences in antibiotic use (DDD per 1000 consultations) according to physician, practice, quality circle (QC), walk-in clinic, and patient characteristics.
Model-estimated differences in antibiotic use | Over 12 months.
  Multilevel regression coefficients estimating differences in antibiotic use (DDD per 1000 consultations) according to physician, practice, QC, walk-in clinic and patient characteristics.
Use of diagnostic tests | Over the ILI season (6 months).
  Number of C-reactive protein (CRP) measurements, blood counts, and chest radiographs per 1000 consultations.
Perceived acceptability of the CRP flowchart | Baseline and after 6 months.
  Perceived acceptability of the CRP flowchart, measured using a French translation of the "Acceptability of Intervention Measure" (5-point Likert scale, higher score means better outcome).
Perceived acceptability of the CRP flowchart assessed by custom questions | Baseline and after 6 months.
  Perceived acceptability of the CRP flowchart, assessed using study-specific custom questions (e.g. "I generally agree with prescribing antibiotics in patients with an acute respiratory infection and a CRP level ≥ 100 mg/L." (question originally asked in French), with answer options according to a 5-point Likert scale, higher scores indicate better outcomes).
Perceived acceptability of shared decision-making | Baseline and after 6 months.
  Perceived acceptability of shared decision-making, measured using a French translation of the "Acceptability of Intervention Measure" (5-point Likert scale, higher score means better outcome).
Perceived acceptability of shared decision-making assessed by custom questions | Baseline and after 6 months.
  Perceived acceptability of shared decision-making, assessed using study-specific custom questions (e.g. "I appreciate the Consultation Support Tool for shared decision-making." (question originally asked in French), with answer options according to a 5-point Likert scale; higher scores indicate better outcomes).
Perceived appropriateness of the CRP flowchart | Baseline and after 6 months.
  Perceived appropriateness of the CRP flowchart, measured using a French translation of "Intervention Appropriateness Measure" (5-point Likert scale, higher score means better outcome).
Perceived appropriateness of the CRP flowchart assessed by custom questions | Baseline and after 6 months.
  Perceived appropriateness of the CRP flowchart, assessed using study-specific custom questions (e.g. "The CRP decision tree corresponds to the patient population in my practice/medical center." (question originally asked in French), with answer options according to a 5-point Likert scale, higher scores indicate better outcomes).
Perceived appropriateness of shared decision-making | Baseline and after 6 months.
  Perceived appropriateness of shared decision-making, measured using a French translation of "Intervention Appropriateness Measure" (5-point Likert scale, higher score means better outcome).
Perceived appropriateness of shared decision-making assessed by custom questions | Baseline and after 6 months.
  Perceived appropriateness of shared decision-making, assessed using study-specific custom questions (e.g. "Shared decision-making in patients with an acute respiratory infection and a CRP level ≥ 50 mg/L and < 100 mg/L corresponds to the patient population in my practice/medical center." (question originally asked in French), with answer options according to a 5-point Likert scale, higher scores indicate better outcomes).
Perceived feasibility of the CRP flowchart | Baseline and after 6 months.
  Perceived feasibility of the CRP flowchart, measured using a French translation of "Feasibility of Intervention Measure" (5-point Likert scale, higher score means better outcome).
Perceived feasibility of the CRP flowchart assessed by custom questions | Baseline and after 6 months.
  Perceived feasibility of the CRP flowchart, assessed using study-specific custom questions (e.g. "CRP testing in patients with an acute respiratory infection can be performed within a reasonable timeframe." (question originally asked in French), with answer options according to a 5-point Likert scale, higher scores indicate better outcomes).
Perceived feasibility of shared decision-making | Baseline and after 6 months.
  Perceived feasibility of shared decision-making, measured using a French translation of "Feasibility of Intervention Measure" (5-point Likert scale).
Perceived feasibility of shared decision-making assessed by custom questions | Baseline and after 6 months.
  Perceived feasibility of shared decision-making, assessed using study-specific custom questions (e.g. "Shared decision-making in patients with an acute respiratory infection and a CRP level ≥ 50 mg/L and < 100 mg/L takes too much time." (question originally asked in French), with answer options according to a 5-point Likert scale, higher scores indicate better outcomes).
Intended adoption of acute respiratory infection guidelines | Baseline and after 6 months.
  Intended adoption of the new ARI guideline using custom questions. Intended adoption of the CRP flowchart using custom questions. Intended adoption of shared decision-making using custom questions.
Fidelity to C-reactive protein | Baseline and after 6 months.
  Fidelity to the CRP flowchart of the new ARI guidelines, using custom questions.
Fidelity to shared decision-making | Baseline and after 6 months.
  Fidelity to shared decision-making of the new ARI guidelines, using custom questions.
Anticipated sustainment of acute repiratory infection guidelines | Baseline and after 6 months.
  Anticipated sustainment of the new ARI guidelines, using custom questions.
Intended adoption of implementation strategies | Baseline and after 6 months.
  Intended adoption of implementation strategies, measured with custom questions (5-point Likert scale, higher score is higher intention to adopt).
Adoption of implementation strategies | Baseline and after 6 months.
  Adoption of implementation strategies, measured with custom questions (single answer, yes/no).
Appropriateness of implementation strategies | Baseline and after 6 months.
  Perceived appropriateness of implementation strategies delivered through and outside QCs, measured with custom questions (5-point Likert scale, higher score is higher appropriateness).
Fidelity in delivering the implementation strategies | During the ILI season (6 months).
  Fidelity of delivering the implementation strategies as intended, using custom questions.
Acceptability of moderator implementation materials | During the ILI season (6 months).
  Acceptability of implementation materials for moderators, measured with the instrument "Acceptability of Intervention Measure" (5-point Likert scale, higher score means better outcome) and additional custom question(s).
Acceptability of physician implementation materials | During the ILI season (6 months).
  Acceptability of implementation materials for physicians, measured with the instrument "Acceptability of Intervention Measure" (5-point Likert scale, higher score means better outcome) and additional custom question(s).
Contextual and individual determinants of adoption | Within 6 months after the ILI season.
  Determinants of adoption of the ARI guidelines identified through qualitative interviews, focus groups, and potentially quantitative data collection.

OTHER OUTCOMES:
Knowledge about acute respiratory infection management | Baseline and after 6 months.
  Knowledge about ARI management according to the new guidelines, measured with a custom questionnaire: "Knowledge questionnaire on the diagnosis and treatment of acute respiratory infections and influenza-like syndromes", (6 questions, of which 3 multiple choice, 3 single choice).
Cost-effectiveness of ARI guideline implementation | Over the ILI season (6 months).
  Incremental cost-effectiveness ratio (ICER), expressed in CHF per percentage point reduction in antibiotic prescribing, comparing the ARI guideline implementation strategy to routine practice.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Mueller, MD, PhD, Principal Investigator — Unisanté, Centre for Primary care and Public Health & University of Lausanne, Switzerland
Locations (1):
- Unisanté, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The non-identifiable data from the physician and moderator surveys, excluding free-text items, will be shared on the institutional data repository data.unisante.ch under the license CC-BY in open access mode. The ownership of these data will be joint between Unisanté and IFIS.
  Billing data cannot be shared due to intellectual property rights and restrictions on reuse of the data.
  Qualitative data from Institute for Implementation Science in Healthcare, University of Zurich (interview data (audio/video files, transcripts)) will not be shared, as the risk of identification remains even after removing names, affiliations and other direct identifiers.
  Non-identifiable quotes of the interview partner, frequencies of codes, or processed/aggregated data will be shared upon reasonable request. These data will not be stored on a data repository as the effort to process data is not considered in proportion to the likelihood that this data will be requested from other research groups.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) from physician questionnaires (excluding free-text responses) will be available via the Unisanté open-access repository starting approximately 12 months after the final data collection (estimated for mid-2027). Data will remain accessible for at least 10 years, after which it will be evaluated for long-term archiving.
Access Criteria: Any researcher will be able to access the non-identifiable IPD from physician questionnaires (excluding free-text) and related documentation via the Unisanté open-data repository. Data will be shared in open and original formats (.csv and others) under a CC-BY license. All other data, including interview materials and SASIS datasets, will not be shared due to confidentiality requirements or legal restrictions.
URL: https://data.unisante.ch/home

REFERENCES:
- [Background] Wolfensberger A, Gendolla SC, Dunaiceva J, Pluss-Suard C, Niquille A, Nicolet A, Marti J, Powell BJ, Naef R, Boillat-Blanco N, Mueller Y, Clack L. Systematic method for developing tailored strategies for implementing point-of-care procalcitonin testing to guide antibiotic prescribing in Swiss primary care: a protocol for a mixed-methods participatory approach. BMJ Open. 2025 Mar 5;15(3):e091285. doi: 10.1136/bmjopen-2024-091285. PMID 40044189
- See also: Description of the study on Unisanté webpage that includes the information sheet for study participants — https://www.unisante.ch/fr/formation-recherche/recherche/projets-etudes/efficacite-implementation-recommandations-nationales
- See also: Description of the project on the website of Swiss National Science Foundation — https://data.snf.ch/grants/grant/212429